CLINICAL TRIAL: NCT02896686
Title: Multicentric, Prospective, Randomized and Simple Blind Study to Determine the Efficacy of the Placement of an Onlay Mesh for Prevention of Incisional Hernia After Loop Ileostomy Closure in Patients With a Prior Rectal Resection for Cancer
Brief Title: Efficacy of an Onlay Mesh for Prevention of Incisional Hernia After Loop Ileostomy Closure
Acronym: ILEOMESH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Aleidis Caro, PhD Aleidis Caro, Hospital Universitari Joan XXIII de Tarragona.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ILEOMESH
Record Dates: First submitted 2016-04-16; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Incisional Hernia
Keywords: Ileostomy closure; Polypropylene Mesh; Incisional hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Abdominal wall closure will be done by continuous polydioxanone (PDS) suture following a SL:WL ratio of 4:1, and the skin will be closed using a subcutaneous purse-string closure
  Interventions: Radiation: Control CT; Other: Clinical Follow Up
- Reinforcement with Mesh (Experimental): Abdominal wall closure will be done by continous polydioxanone (PDS) suture following a SL:WL ratio of 4:1.
  The incision is reinforced with onlay placement of a light polypropylene mesh (3 cm wide and the length corresponding to the incision), fixed to the aponeurosis with interrupted polyglactin (Vycril) suture.
  The skin will be closed using a subcutaneous purse-string closure
  Interventions: Radiation: Control CT; Other: Clinical Follow Up; Procedure: Reinforcement with Light Polypropylene Mesh

INTERVENTIONS:
Radiation: Control CT — At the end of the follow up (12 Months) a CT scan will be done. Radiologically the incisional hernia is defined as a solution of continuity of the abdominal wall seen on the abdominal CT scan with the patient at rest.
  The radiologist is blinded to the patient's history and the technique used for fascial closure.
Other: Clinical Follow Up — The presence of incisional hernia was evaluated by physical examination at scheduled clinical visits (3 and 6 months after surgery) Clinically, an incisional hernia is defined as the presence of a reducible bulge or protrusion at the laparotomy incision scar, palpable during the Valsalva maneuver.
Procedure: Reinforcement with Light Polypropylene Mesh — Reinforcement with Light Polypropylene Mesh
  Arms: Reinforcement with Mesh

SUMMARY:
The aim of the present study is to determine the efficacy of the placement of an onlay mesh to prevent incisional hernia after loop ileostomy closure in patients with a prior rectal resection for cancer

DETAILED DESCRIPTION:
The primary aim of the study is to determine the efficacy of the placement of an onlay mesh for prevention of incisional hernia after loop ileostomy closure in patients with a prior rectal resection for cancer. The efficacy will be evaluated by physical examination 3, 6 and 12 months after surgery and by abdominal CT scan one year after stoma closure.

Secondary aims are to evaluate the tolerability and safety of the prothesis; complications, quality of life and the need for further treatments will be compared between the groups.

This is a multicentric study that will include patients operated on in hospitals in Catalunya for loop ileostomy closure after a prior rectal resection for rectal cancer. Elective surgery for loop ileostomy closure with ASA<4. Exclusion criteria include patients with allergy or intolerance to polypropilene, with a prior mesh on the abdominal wall, ASA ≥IV, patients with a life expectancy of <12 months, chronic renal failure in haemodialysis and patients on steroid therapy.

Patients that agree to participate in the study will be randomized using an electronic formula (Excel) of a uniformly distributed variable assigning case/control randomly until the total number of patients are included.

In the control group, after the digestive tract is reconstructed, the closure of the abdominal wall will be performed with a continuous suture of PDS loop 1/0 following Jenkins 4:1 rule and the skin will be closed using a subcutaneous purse-string closure. Patients in the study group will have the same procedure performed, and after the aponeurosis closure with PDS loop, an onlay light polypropilene mesh will be placed.

Each participant will have an assigned code depending on the participating Centre that will maintain anonymity at all times. All of the information will be registered in a database specifically designed for the study.

Statistical analysis will be performed by a descriptive study of the demographic variables and the incidence of incisional hernia after loop ileostomy closure. A comparative study between the groups will be performed using X2 test for categorical variables and t Student test or U-Mann for continuous variables. A binary logistic regression will also be performed to analyse the influence of each variable and to predict if the interventions produce incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

* patients operated on in hospitals in Catalunya for loop ileostomy closure after a prior rectal resection for rectal cancer.
* elective surgery for loop ileostomy closure
* ASA (American Society of Anesthesiologists)<4

Exclusion Criteria:

* allergy or intolerance to polypropilene
* patients with a prior mesh on the abdominal wall
* ASA ≥IV
* patients with a life expectancy of <12 months
* chronic renal failure in haemodialysis
* patients on steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 12 months
  The primary endpoint is the incidence of incisional hernia, either symptomatic or asymptomatic in the mesh and suture-only groups. Because appearance of an incisional hernia occurs within the first months after laparotomy, assessment of efficacy was carried out during scheduled clinical visits over a period of 12 months. The presence of incisional hernia was evaluated by physical examination at scheduled clinical visits and radiologically by an abdominal CT scan performed at the end of follow-up (6 months after operation).

SECONDARY OUTCOMES:
Perioperative complications | 30 days
  Secondary endpoints are perioperative complications, including wound infection, hematoma, pain and reoperation.
Quality of life of the patients | 3, 6 and 12 months after surgery
  The quality of life was evaluated by the SF-36 Quality of life test, during scheduled clinical visits over a period of 12 months.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://cirurgiahj23.wordpress.com